CLINICAL TRIAL: NCT06086756
Title: The Influence of Mood on Response to Virtual Reality-Based Exposure for Public Speaking Anxiety
Brief Title: Virtual Reality Intervention for Speech Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7164E
Record Dates: First submitted 2023-10-02; First posted 2023-10-17 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Public Speaking; Speech Anxiety
MeSH Terms: conditions — Speech; Glossophobia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Mood Induction via positive film clips (Experimental): The standardized procedures outlined in our laboratory's previously conducted study (Stathopoulou, Pollack, & Otto, 2018) will be followed. Participants will be presented with two brief film clips on a computer monitor or TV screen. These film clips were selected to elicit positive affect. As utilized in past lab study procedures, participants will be asked to: "Let yourself experience whatever emotions you have, as fully as you can. Don't try to hold back, or hold in, your feelings" (Stathopoulou, Pollack, & Otto, 2018). Together, the two film clips will last for approximately 5 minutes.
  Interventions: Behavioral: Exposure intervention plus positive mood induction
- Negative Mood Induction via negative film clips (Experimental): The standardized procedures outlined in our laboratory's previously conducted study (Stathopoulou, Pollack, & Otto, 2018) will be followed. Participants will be presented with two brief film clips on a computer monitor or TV screen. These film clips were selected to elicit negative affect. As utilized in past lab study procedures, participants will be asked to: "Let yourself experience whatever emotions you have, as fully as you can. Don't try to hold back, or hold in, your feelings" (Stathopoulou, Pollack, & Otto, 2018). Together, the two film clips will last for approximately 5 minutes.
  Interventions: Behavioral: Exposure intervention plus negative mood induction

INTERVENTIONS:
Behavioral: Exposure intervention plus positive mood induction — Positive mood induction followed by a brief VR exposure session for public speaking anxiety.
  Arms: Positive Mood Induction via positive film clips
Behavioral: Exposure intervention plus negative mood induction — Negative mood induction followed by a brief VR exposure session for public speaking anxiety.
  Arms: Negative Mood Induction via negative film clips

SUMMARY:
Exposure-based cognitive behavior therapy is an efficacious treatment for speech anxiety and has been delivered effectively in a virtual reality (VR) environment. The present study is designed to evaluate whether mood state moderates outcome to a brief VR exposure intervention.

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare outcomes of VR exposure therapy for college students with public speaking anxiety following a positive or negative mood induction. The overarching aim of the present study is to determine whether mood state prior to engaging in a brief VR exposure therapy session for public speaking anxiety impacts treatment outcomes.

The study involves three phases: (1) initial screening, (2) in-person assessment and brief exposure intervention for a subset of participants with elevated public speaking anxiety, and (3) a one-week follow-up assessment conducted online. Students who choose to participate and screen high on a public speaking anxiety scale will be assigned to a positive or negative mood induction condition prior to undergoing VR based exposure therapy. Public speaking and social anxiety outcomes are measured immediately post-intervention and one week later.

Researchers will compare participants given a positive mood induction to participants given a negative mood induction to see if public speaking anxiety outcomes differ.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of 18 years of age or older
* Current student at Boston University
* Ability to read English to provide informed consent
* Familiarity with a computer keyboard and mouse or a touch screen device (e.g. phone, tablet).
* For Phase 2: speech anxiety scale score of ≥ 14 on the Personal Report of Communication Apprehension, Public Speaking Subscale (PRCA-PS)

Exclusion Criteria:

* Previous participation (i.e., no participant may take the survey more than once).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Public Speaking Anxiety | Comparison of pre-exposure scores to scores from post-treatment, approximately 2 week post-screen
  Assessed using the Personal Report of Communication Apprehension, Public Speaking Subscale (PRCA-PS)

SECONDARY OUTCOMES:
Valence | Comparison of pre-exposure scores to scores from follow up survey, 1 week post-exposure
  Self-report measure of how participant feels about having to give a speech
Social Phobia | Comparison of pre-exposure scores to scores from follow up survey, 1 week post-exposure
  Assessed using the social phobia inventory (SPIN)
Public Speaking Anxiety | Comparison of pre-exposure scores to scores from follow up survey, 1 week post-exposure
  Assessed using the PRCA-PS

CONTACTS AND LOCATIONS:
Overall Officials: Elias Culver, Principal Investigator — Boston University
Locations (1):
- Center for Anxiety and Related Disorders, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No